CLINICAL TRIAL: NCT03876847
Title: Genetics of Spontaneous Coronary Artery Dissection (SCAD-INSPIRE Genetics): A Substudy of the INSPIRE Registry
Brief Title: Genetics of Spontaneous Coronary Artery Dissection (SCAD-INSPIRE Genetics)
Acronym: SCAD-INSPIRE
Status: Enrolling by invitation | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050343
Record Dates: First submitted 2019-02-04; First posted 2019-03-15 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva, buccal swab, or blood sample kit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous Coronary Artery Disection: The spontaneous coronary artery disection (SCAD) diagnosis will be based on independent review of clinical presentation, cardiac imaging, and angiography findings by three cardiologists. The determination will be evidence of linear luminal defect (intimal flap) detection, luminal narrowing or occlusion confirmed to be a dissection on further imaging, or by clinical judgment classifying it as definite SCAD.
- Control: A set of controls will be used for genetic analysis. These controls will pulled from subjects in the INSPIRE registry that had coronary angiography at Intermountain Medical Center for stable angina and meet inclusion/exclusion criteria.

SUMMARY:
Spontaneous coronary artery dissection (SCAD) is a rare cause of coronary ischemia and infarction where a tear in blood vessel wall either restricts the flow of blood or the blood becomes trapped in between the layers of the vessel causing the vessel to impinge on the lumen and causing an obstruction or restriction of blood flow. The ultimate goal of this proposal is to further understand the risk factors leading to SCAD with a focus on familial and genetic causes of SCAD.

DETAILED DESCRIPTION:
For this study, we will ascertain clinical data and biological samples from a cohort of SCAD patients identified using retrospective review of medical records and prospective surveillance of Intermountain patients that undergo coronary angiography. The SCAD diagnosis will be based on independent review of clinical presentation, cardiac imaging, and angiography findings by two cardiologists and a third cardiologist in case of disagreement. It is anticipated that we hope to recruit 100 SCAD patients.

Enrollment of these subjects will be done under the INSPIRE registry. The subjects will be asked to sign a consent, provide biological samples, and complete questionnaires related to SCAD as part of the INSPIRE registry.

The SCAD cases will be matched to records in the Intermountain Genealogy Registry (IGR) to allow for the identification of possible high-risk SCAD families. Risk of first and second degree relatives will also be assessed. The obtained blood samples will be processed, stored and genotyped.

ELIGIBILITY:
Inclusion Criteria:

SCAD Cases

1. Subjects of all ages, gender, or race
2. Subjects had coronary angiography.
3. Subjects had suspected SCAD as based on clinical report.

Controls

1. INSPIRE subject that had coronary angiography at Intermountain Healthcare for stable angina.
2. Subjects had no or mild atherosclerotic heart disease at time of angiography.
3. Age at last visit as recorded in the Intermountain EDW at least 50 years or older.
4. Not screened as possibly having a SCAD or coronary artery dissection diagnosis.

Exclusion Criteria:

SCAD Cases

1. Independent review of cardiac imaging and clinical presentation by three cardiologists determine the coronary angiography was not a result of SCAD.
2. Imaging from time of coronary angiography of poor quality as to not allow for proper determination of SCAD.
3. Inability to determine criteria as outlined above.
4. Subjects that have had a heart transplant.
5. Subjects that have had a bone marrow transplant.
6. Inability or refusal of the patient and/or the patient's legally acceptable representative to provide informed consent or blood sample for any reason.
7. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the trial.

Controls

1. Subjects that have a heart transplant.
2. Subjects that have a bone marrow transplant.
3. Subjects with any of the following diagnosis at anytime

   1. Heart failure
   2. Heart valve disease
   3. Thoracic aortic aneurysm and dissection
   4. Ehlers-Danlos syndrome
   5. Shprintzen-Goldberg syndrome
   6. Marfan syndrome
   7. Loeys-Dietz aortic aneurysm syndrome
   8. Arterial tortuosity syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be Intermountain Healthcare patients. The case subjects will be SCAD patients and the control population for the genetics will be Intermountain angiography patients without SCAD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-17 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic variants | at enrollment
  To determine genetic variants among spontaneous coronary artery dissection (SCAD) patients, we will do genotyping including target sequencing and whole exome/genome sequencing on samples provided by SCAD patients. The primary focus of this sequencing will be to determine rates of variants in genes that cause cardiac-related connective tissue disorders.